CLINICAL TRIAL: NCT06621732
Title: Combating the Diagnostic Impasse in Mitochondrial Diseases: a Transcriptomic Approach in Fibroblasts and Blood Cells
Acronym: RNAseq
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-AOIP-07
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitochondrial disease (Experimental)
  Interventions: Procedure: cutanous biopsy and blood sample

INTERVENTIONS:
Procedure: cutanous biopsy and blood sample — cutanous biopsy and blood sample

SUMMARY:
Next-generation sequencing (NGS), and in particular whole exome sequencing (WES) or genome sequencing (WGS), has enabled a significant technical advance that has considerably improved genetic diagnostics. However, around 50% of patients still remain undiagnosed and are in diagnostic limbo. One of the causes of this is pathogenic variants that modify transcript expression and/or RNA splicing. These variants may be located in deep intronic or intergenic regions, or in the coding sequence, synonymous or missense variants, also having pathogenic consequences on splicing or gene expression. It is very often difficult to interpret the pathogenicity of these variants, which often remain variants of uncertain significance (VSI). The usefulness of transcriptome sequencing (RNA-seq) in the genetic diagnosis of MM has been demonstrated in recent years by several teams with diagnostic yields of 10% to 35%. These studies are ideally performed using muscle tissue, as MMs are most often expressed in tissues with high energy metabolism such as muscle, heart, brain or liver. However, as biopsies of these tissues are difficult to obtain, most transcript studies are performed using fibroblasts obtained from skin biopsies. Indeed, extreme regulatory defects such as loss of expression or aberrant splicing can be detected in fibroblasts, even though the physiological consequence on fibroblasts may be negligible. However, some patients also refuse these biopsies and may remain in diagnostic limbo in the absence of functional analysis to confirm the pathogenicity of the variants identified. RNA studies can also be performed using RNA extracted from blood cells on PAXGene tubes. The quantity of RNA extracted is lower than that extracted from fibroblasts, but this type of analysis avoids a more invasive procedure, saves technical time by avoiding the manips associated with cell culture, and saves time for the patient by enabling immediate extraction from the blood tube without waiting for cell culture. Frésard et al showed in patients with 16 different Mendelian pathologies that RNA-seq on blood cells identified a diagnosis in 7.5% of patients tested. Their approach revealed both expression variations and splicing anomalies.

The investigators therefore propose to carry out a transcript study using high-throughput RNA sequencing (RNA-Seq), in parallel on RNA extracted from fibroblasts and on RNA extracted from blood cells, on 10 patients with suspected mitochondrial disease in whom variants of uncertain significance in candidate genes (VSI+) have been identified.

The investigators chose to target our study on patients with VSI+, previously identified by NGS, to facilitate interpretation of the RNA-Seq data within the framework of a "pilot" study. In these patients, who carry variants in candidate genes, the investigators will focus our bioinformatics analysis on these genes. For the interpretation of VSI+, a targeted approach using Sanger sequencing based on RT-PCR, or quantification of gene expression using quantitative PCR, is also feasible, but requires custom development for each variant, which is very time-consuming and not insignificantly expensive. The advantage of an RNA-seq approach is that it homogenizes the diagnostic strategy for patients, saves analysis time and therefore reduces the time spent in diagnostic wandering. Finally, the drastic reduction in the cost of NGS sequencing means that this technique could be used routinely as a complement to exome/genome sequencing. It could therefore eventually be applied not only to patients with VSI+ but also, in the absence of evidence of potentially pathogenic variants, as an aid to filtering variants identified by WES/WGS.

ELIGIBILITY:
Inclusion Criteria:

General criteria: major or minor patients, sporadic or isolated cases

* Pathology-related criteria :

  * Patients with suspected mitochondrial disease according to Morava criteria
  * Identification of a predicted VSI, "possibly pathogenic" by SPICE and/or SpliceAI biοstatistical and biοinfοrmatic prediction tools, in a gene :
* Compatible with the patient's phenotype
* With sufficient expression in blood (TPM>1, GTEX) predicted as "possibly pathogenic" by SPICE and/or SpliceAI biοstatistical and biοinfοrmatic prediction tools.
* Signature of informed consent, for minor patients signature of at least one of the 2 parents or the representative of parental authority

Exclusion Criteria:

* Patient whose identified VSI is in the same gene as a patient already included in the study;
* Persons deprived of liberty by judicial or administrative decision;
* Persons hospitalized without consent;
* Persons of full age or minors under legal protection or unable to express their consent;
* Inability of the subject to cooperate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The main objective is to establish whether the study of transcripts from RNA extracted from blood cells yields the same results as a study carried out using RNA extracted from fibroblasts in patients with mitochondrial diseases. | inclusion visit
  Concordance of results on fibroblasts and blood cells for 100% of variants studied.

SECONDARY OUTCOMES:
Establish a definitive diagnosis in these patients with diagnostic impasses. | 17 months
  Number of patients for whom the 2 techniques led to a definitive diagnosis, i.e. reclassification of "variants of undetermined significance" as "pathogenic variants".
Test our ability to analyze RNA-Seq data. | 17 months
  Concordance of results with the data analysis tool Galiléo (Integragen) and a "home-made" pipeline in collaboration with bio-informaticians from the Maison de la Modélisation, Simulation et Interaction, Université Côte d'Azur/CHU de Nice.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de NIce, Nice, Alpes-maritimes
  - CHU de Montpellier, Montpellier